CLINICAL TRIAL: NCT00001189
Title: The Treatment of Grade I Sarcomas and Benign, Non-Metastasizing Highly Invasive Soft Tissue Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 830227; 83-C-0227
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-05

CONDITIONS: Sarcoma; Neoplasms
Keywords: Adjuvant Radiotherapy; Low-Grade Sarcoma; Radiotherapy; Randomized Study; Sarcoma; Surgery
MeSH Terms: conditions — Sarcoma; Neoplasms | interventions — Radiotherapy

INTERVENTIONS:
Procedure: radiotherapy

SUMMARY:
Patients with Grade I soft tissue sarcomas or benign, non-metastasizing invasive soft tissue tumors will receive wide local excision and be prospectively randomized as to either receive or not receive radiation therapy.

DETAILED DESCRIPTION:
This is a randomized study. Patients undergo surgical excision of all gross disease and then are randomized to Arm I or Arm II.

Arm I: Radiotherapy. Involved-field irradiation.

Arm II: No further treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Biopsy-proven grade I soft tissue sarcoma or one of the following benign but highly invasive soft tissue tumors:

Abdominal and extra-abdominal fibromatosis (desmoid,

aggressive fibromatosis),

Dermatofibrosarcoma protuberans,

Intramuscular lipoma (infiltrating lipoma),

Diffuse lipomatosis,

Leiomyoma of deep soft tissue,

Diffuse giant cell tumor of tendon sheath (proliferative synovitis).

No clinical evidence of metastases in regional nodes or more distant sites.

No primary intraperitoneal or retroperitoneal tumors.

Resection of all gross tumor at the time of surgical excision required (margins may be pathologically positive or negative).

No von Recklinghausen's disease.

PRIOR/CONCURRENT THERAPY:

Biologic Therapy: Not specified.

Chemotherapy: No prior chemotherapy for sarcoma.

Endocrine Therapy: Not specified.

Radiotherapy: No prior radiotherapy for sarcoma.

Surgery: No more than 4 months since definitive surgery for

primary lesion or recurrence.

No prior amputation.

PATIENT CHARACTERISTICS:

Age: 18 and over.

Performance status: Not specified.

Hematopoietic: Not specified.

Hepatic: No cirrhosis.

Renal: No evidence of severe renal impairment.

Cardiovascular: No ischemic heart disease.

OTHER:

No prior malignancy except basal cell carcinoma.

No serious infection.

No active bleeding disorder.

No severe concomitant disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1983-12; Study Completion 2001-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Wara WM, Phillips TL, Hill DR, Bovill E Jr, Luk KH, Lichter AS, Leibel SA. Desmoid tumors--treatment and prognosis. Radiology. 1977 Jul;124(1):225-6. doi: 10.1148/124.1.225. PMID 405711